CLINICAL TRIAL: NCT04724369
Title: A Prospective Phase 3 Multi-center Study to Assess the Efficacy and Safety of 18F-mFBG PET Imaging in Subjects with Neuroblastoma
Brief Title: Open-Label Study of 18F-mFBG for Imaging Neuroblastoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Innervate Radiopharmaceuticals LLC (Formerly: Illumina Radiopharmaceuticals LLC) (Industry)
Collaborators: New Approaches to Neuroblastoma Therapy Consortium (Other); Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRP101-301
Record Dates: First submitted 2021-01-18; First posted 2021-01-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-01

CONDITIONS: Neuroblastoma
Keywords: 18F-mFBG; meta-fluorobenzylguanidine
MeSH Terms: conditions — Neuroblastoma | interventions — 3-fluorobenzylguanidine

STUDY DESIGN:
Intervention Model Description: Comparison of PET imaging interpretation and expert assessment for presence or absence of neuroblastoma tumor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study Cohort: Subjects with known or presumed neuroblastoma (Experimental): Drug: 18F-mFBG Positron-emitting radiopharmaceutical 18F-mFBG as an imaging agent for identification of neuroblastoma.
  Other Names:
  * meta-fluorobenzylguanidine
  * IRP101
  Interventions: Drug: 18F-MFBG

INTERVENTIONS:
Drug: 18F-MFBG — Positron-emitting tomography (PET) (either PET/CT or PET/MR) imaging agent
  Other Names: meta-fluorobenzylguanidine; IRP101

SUMMARY:
This is a Phase 3 study evaluating the positron-emitting radiopharmaceutical 18F-mFBG as an imaging agent for confirming or excluding the presence of neuroblastoma

DETAILED DESCRIPTION:
This is a prospective, Phase 3, multi-center, open-label study designed to assess the use of 18F-mFBG PET imaging in subjects with known or presumed neuroblastoma. Eligible participants will have either histopathologically established diagnosis of neuroblastoma or a presumed diagnosis based on signs, symptoms, physical examination, imaging findings, and laboratory and genetic test results.

Subjects will only be administered 18F-mFBG if they have undergone or are scheduled to undergo a 123I-mIBG or 18F-FDG scan within 30 days of the date of the 18F-mFBG scan. Subjects should not have received any chemotherapy, immunotherapy or radiotherapy between the clinical and 18F-mFBG imaging studies.

18F-mFBG PET studies and clinical 123I-mIBG scans will be evaluated off-site by 3 independent radiologists and/or nuclear medicine physicians who are blinded to all subject information. Blinded readers will record whether findings on 18F-mFBG and 123I-mIBG scans are consistent with presence of neuroblastoma (Disease +) or absence of disease (Disease -).

Subject-level diagnostic performance will be assessed on the basis of positive and negative percent agreement (PPA and NPA) between the blinded 18F-mFBG scan interpretations and disease status (+ or - for neuroblastoma) as independently assessed by an Expert Panel of pediatric oncologists.

Secondary efficacy analyses will compare PPA and NPA between 18F-mFBG and 123I-mIBG interpretations provided by the blinded readers.

ELIGIBILITY:
Inclusion Criteria:

1. a) An established diagnosis of neuroblastoma based on unequivocal histopathology from tissue obtained at any time prior to enrolment in the trial; OR b) A presumed diagnosis of neuroblastoma based on signs, symptoms, physical examination, imaging findings, and laboratory and genetic test results, including individuals in whom therapy has already been empirically initiated.
2. The subject has undergone or is scheduled to undergo evaluation of neuroblastoma disease status, including at least one functional imaging study (123I-mIBG or 18F-FDG), within 30 days prior to the date of 18F-mFBG imaging, with no interval therapy between such evaluation and investigational drug administration.
3. Ability of subject or subject's legal guardian to understand and sign a written informed consent document, including, for subjects age 7-17, an assent form.

Exclusion Criteria:

1. The subject was previously entered into this study.
2. The subject is pregnant, breast feeding, or menarchal and unwilling to use effective contraception during the study.
3. The subject has a history or suspicion of significant allergic reaction or anaphylaxis to any components of the 18F-mFBG imaging agent.
4. The subject is unable to lie flat or remain still for approximately 30 minutes to allow performance of a PET scan.
5. The subject uses medications that are known to interfere with uptake of NET-dependent agents and these medications cannot be safely withheld 24 hours before study procedures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
PET Scan Identification of Neuroblastoma | Imaging at 60 minutes
  Focal 18F-mFBG uptake (presence or absence) when imaging at 60 minutes with PET/CT or PET/MR, reported as positive and negative predictive agreement with expert oncologist assessment for presence of neuroblastoma

SECONDARY OUTCOMES:
Comparison of 18F-mFBG PET With Clinical 123I-mIBG Imaging | Scan interpretation up to one month after intervention.
  This objective will be assessed using the secondary endpoint of focal increased 123I-mIBG uptake (presence or absence), reported as positive and negative predictive agreement with expert oncologist assessment for presence of neuroblastoma
Number of subjects with adverse events graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE), Version 5. | 24 hours following 18F-mFBG administration.
  Description: Assessments based on changes between pre- and post-18F-mFBG administration physical examination findings, vital signs measurements, blood test results including hematology and biochemistry, and electrocardiograms (ECGs).

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Riley Hospital for Children - Indiana University, Indianapolis, Indiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No